CLINICAL TRIAL: NCT03660839
Title: A Randomized, Open Label, Parallel-group, Single Dose Regimen, Phase 2a Study, to Investigate the Clinical and Parasiticidal Activity and the Pharmacokinetics of 3 Dose Levels of Artefenomel (OZ439) Given in Combination With Ferroquine (FQ) and FQ Alone, in African Patients With Uncomplicated Plasmodium Falciparum Malaria
Brief Title: Study to Investigate the Clinical and Parasiticidal Activity and Pharmacokinetics of Different Doses of Artefenomel and Ferroquine in Patients With Uncomplicated Plasmodium Falciparum Malaria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Medicines for Malaria Venture (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACT14655; U1111-1191-5573 (Other: UTN)
Record Dates: First submitted 2018-08-20; First posted 2018-09-07 (Actual); Results first posted 2020-12-02 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Plasmodium Falciparum Infection
MeSH Terms: interventions — artefenomel; ferroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Ferroquine 400 milligram (mg) (Experimental): On Day 0, participants received orally a single dose of FQ 400 mg (4 capsules of 100 mg) in fasted condition.
  Interventions: Drug: Ferroquine (SSR97193)
- Ferroquine 400 mg + Artefenomel 300 mg (Experimental): On Day 0, participants received orally a single dose of FQ 400 mg (4 capsules of 100 mg) in fasted condition followed by OZ439 300 mg oral suspension.
  Interventions: Drug: Artefenomel (OZ439); Drug: Ferroquine (SSR97193)
- Ferroquine 400 mg + Artefenomel 600 mg (Experimental): On Day 0, participants received orally a single dose of FQ 400 mg (4 capsules of 100 mg) in fasted condition followed by OZ439 600 mg oral suspension.
  Interventions: Drug: Artefenomel (OZ439); Drug: Ferroquine (SSR97193)
- Ferroquine 400 mg + Artefenomel 1000 mg (Experimental): On Day 0, participants received orally a single dose of FQ 400 mg (4 capsules of 100 mg) in fasted condition followed by OZ439 1000 mg oral suspension.
  Interventions: Drug: Artefenomel (OZ439); Drug: Ferroquine (SSR97193)

INTERVENTIONS:
Drug: Artefenomel (OZ439) — Pharmaceutical form: Granules for oral suspension Route of administration: Oral
  Arms: Ferroquine 400 mg + Artefenomel 1000 mg; Ferroquine 400 mg + Artefenomel 300 mg; Ferroquine 400 mg + Artefenomel 600 mg
Drug: Ferroquine (SSR97193) — Pharmaceutical form: Capsule Route of administration: Oral

SUMMARY:
Primary Objective:

To show the contribution of artefenomel (OZ439) to the clinical and parasiticidal effect of OZ439/Ferroquine (FQ) combination by analyzing exposure-response of OZ439 measured by Day 28 polymerase chain reaction (PCR)-corrected adequate clinical and parasitological response (ACPR) for the effect and the area under the curve (AUC) of OZ439 as pharmacokinetic (PK) predictor.

Secondary Objectives:

* To evaluate the exposure-response of OZ439 combined with FQ on crude Day 28 ACPR.
* To evaluate the dose response of OZ439 combined with FQ on PCR-corrected and crude Day 28 ACPR.
* To evaluate the dose-response of OZ439 combined with FQ on selected secondary endpoints.
* To evaluate the safety and tolerability of different dosages of OZ439 in combination with FQ and FQ alone.
* To characterize the PK of OZ439 in plasma, and of FQ and its active metabolite SSR97213 in blood.

DETAILED DESCRIPTION:
The duration of the study was up to 32 days, including up to 1 day screening period before the single-dose treatment, 5 days of post-treatment surveillance (included 2 to 4 days hospitalization) and 24±2 days follow-up period.

ELIGIBILITY:
Inclusion criteria :

Participants (14-69 years old inclusive) with body weight within 35 and 90 kilograms (kg), with uncomplicated Plasmodium falciparum (P. falciparum) malaria, with a fever as defined with axillary temperature greater than or equal to (>=) 37.5 degree Celsius (°C) or oral/ rectal/ tympanic temperature >=38°C or history of fever in the previous 24 hours (history of fever was documented), with a mono-infection with P. falciparum and parasitemia (microscopically, blood smear) >= 3,000 and less than or equal to (<=) 50,000 asexual parasites per microliter of blood.

Exclusion criteria:

* Presence of severe malaria.
* Known history or evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, respiratory, endocrine, immunological, infectious, neurological (in particular convulsions), malignancy, psychiatric disease or symptoms which, in the judgment of the investigator, might confuse the interpretation of the safety information.
* Severe vomiting defined as more than 3 times in the 24 hours prior to enrollment in the study or inability to tolerate oral treatment or severe diarrhea defined as 3 or more watery stools per day.
* Severe malnutrition defined as a body mass index of less than 16 kg per meter square for adults and for children Z-score less than (<) -3 or weight for age (%) of the median <60.
* Splenectomized participants or presence of surgical scar on left hypochondrium.
* Known history of hypersensitivity, allergic, or anaphylactoid reactions to FQ or other amino quinolines or to OZ439 or OZ277 or any of the excipients.
* Participant treated with anti-malarial treatment:
* With piperaquine phosphate-based compound, mefloquine, naphthoquine or sulphadoxine/pyrimethamine within the previous 6 weeks.
* With amodiaquine or chloroquine within the previous 4 weeks.
* With quinine, halofantrine, lumefantrine-based compounds and any other anti-malarial treatment or antibiotics with antimalarial activity (including cotrimoxazole, tetracyclines, quinolones and fluoroquinolones, and azithromycin) within the past 14 days.
* With any herbal products or traditional medicines, within the past 7 days.
* Previous treatment within 5 times the half-life or within the last 14 days, whichever the longest, which were: strong Cytochrome P450 (CYP) 2C or CYP3A inhibitors and/or moderate inhibitors but inhibiting both CYP2C and CYP3A and/or CYP inducers.
* Any treatment known to induce a prolongation of QT interval.
* Participated in any trial investigating OZ439 and/or FQ compounds.
* Previous participation in any malaria vaccine study or received malaria vaccine in any other circumstance.
* Enrolled in another clinical trial within the past 4 weeks or during the study period.
* Mixed Plasmodium infection.
* Presence of Hepatitis A - immunoglobulin, Hepatitis B surface antigen or Hepatitis C virus antibody and/or known to had active Hepatitis C virus ribonucleic acid.
* Laboratory parameters with abnormalities deemed clinically significant by the investigator.
* Abnormal Liver Function Test: aspartate transferase greater than (>) 2 upper limit of normal range (ULN), or alanine transferase >2 ULN or total bilirubin >1.5 ULN.
* Positive pregnancy test at study screening for female participants of childbearing potential.
* QT interval corrected using Fridericia formula (QTcF) >450 milliseconds at screening or pre-dose.
* Hypokalemia (<3.5 millimoles per liter [mmol/L]), hypocalcemia (<2.0 mmol/L) or hypomagnesemia (<0.5 mmol/L) at screening or pre-dose.
* Family history of sudden death or of congenital prolongation of the QT interval or known congenital prolongation of the QT-interval or any clinical condition known to prolong the QT interval e.g., participants with a history of symptomatic cardiac arrhythmias including atrial fibrillation or with clinically relevant bradycardia.
* Participant not suitable for participation, whatever the reason, as judged by the Investigator, included medical or clinical conditions, or participants potentially at risk of noncompliance to study procedures or unable to drink.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 14 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2018-09-11 (Actual); Primary Completion 2019-11-06 (Actual); Study Completion 2019-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (7):
- Investigational Site Number 2040001, Cotonou, Benin
- Burkina Faso (2):
  - Investigational Site Number 8540002, Banfora
  - Investigational Site Number 8540001, Ouagadougou
- Gabon (2):
  - Investigational Site Number 2660002, Lambaréné
  - Investigational Site Number 2660001, Libreville
- Investigational Site Number 4040002, Siaya, Kenya
- Investigational Site Number 8000001, Tororo, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Gansane A, Lingani M, Yeka A, Nahum A, Bouyou-Akotet M, Mombo-Ngoma G, Kaguthi G, Barcelo C, Laurijssens B, Cantalloube C, Macintyre F, Djeriou E, Jessel A, Bejuit R, Demarest H, Marrast AC, Debe S, Tinto H, Kibuuka A, Nahum D, Mawili-Mboumba DP, Zoleko-Manego R, Mugenya I, Olewe F, Duparc S, Ogutu B. Randomized, open-label, phase 2a study to evaluate the contribution of artefenomel to the clinical and parasiticidal activity of artefenomel plus ferroquine in African patients with uncomplicated Plasmodium falciparum malaria. Malar J. 2023 Jan 3;22(1):2. doi: 10.1186/s12936-022-04420-2. PMID 36597076

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 7 active sites in 5 countries. Total of 448 participants were screened between 11 September 2018 and 09 October 2019, of which 140 were randomized to 1 of 4 treatment arms and those who failed to meet inclusion criteria were considered as screen failure.
Pre-assignment Details: All eligible participants were randomized via a centralized randomization system using interactive response technology to 1 of the 4 arms in 1:1:1:1 ratio. Day 0 (drug administration day, per protocol) was considered as Day 1 for all analysis using Safety population as per Clinical Data Interchange Standards Consortium convention.
Groups:
- Ferroquine (FQ) 400 Milligram (mg): On Day 0, participants received orally a single dose of FQ 400 mg (4 capsules of 100 mg) in fasted condition.
- Ferroquine 400 mg + Artefenomel (OZ439) 300 mg: On Day 0, participants received orally a single dose of FQ 400 mg (4 capsules of 100 mg) in fasted condition followed by OZ439 300 mg oral suspension.
Period: Overall Study
Arm/Group | Ferroquine (FQ) 400 Milligram (mg) | Ferroquine 400 mg + Artefenomel (OZ439) 300 mg | Ferroquine 400 mg + Artefenomel 600 mg | Ferroquine 400 mg + Artefenomel 1000 mg
Started | 35 | 36 | 36 | 33
Completed (Completed study treatment.) | 35 | 36 | 36 | 33
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all randomized participants.
Groups:
- Ferroquine 400 mg: On Day 0, participants received orally a single dose of FQ 400 mg (4 capsules of 100 mg) in fasted condition.
- Total: Total of all reporting groups
Arm/Group | Ferroquine 400 mg | Ferroquine 400 mg + Artefenomel 300 mg | Ferroquine 400 mg + Artefenomel 600 mg | Ferroquine 400 mg + Artefenomel 1000 mg | Total
Number analyzed (Participants) | 35 | 36 | 36 | 33 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.4 (13.20) | 21.8 (11.49) | 20.7 (8.57) | 22.2 (11.28) | 22.5 (11.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 28 | 26 | 20 | 97
  Male | 12 | 8 | 10 | 13 | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 35 | 36 | 35 | 33 | 139
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Polymerase Chain Reaction (PCR)-Corrected Adequate Clinical and Parasitological Response (ACPR) at Day 28 (ACPR28)
Description: ACPR:absence of parasitemia at Day 28, irrespective of axillary temperature(AT), participants not meeting any criteria of early therapy failure(ETF):Danger signs(DS)/symptoms of complicated(SoC)/severe malaria(SM) at Day 1, 2 or 3 in presence of parasitemia, concomitant to at least 1 positive parasitemia;or parasitemia on Day 2 >Day 0 irrespective of AT;or parasitemia on Day 3 with AT>=37.5 degree Celsius (°C);or parasitemia count on Day 3 >=25 percent (%) on Day 0, or late clinical failure (LCF):DS/SM in presence of parasitemia between Day 4 and 28,concomitant to at least one positive parasitemia;or presence of parasitemia and AT>=37.5°C on Day 4 to Day 28, or late parasitological failure(LPF):presence of parasitemia between Day 7 and 28 and AT<37.5°C and without rescue therapy. PCR-corrected ACPR applied to recrudescence (appearance of asexual parasites after clearance of initial infection with genotype identical to that present at Baseline), excluding participants with reinfection.
Time Frame: Day 28
Population: Pharmacokinetic/Pharmacodynamic (PK/PD) efficacy population: who received at least 1 dose of OZ439/FQ with parasitologically confirmed Plasmodium falciparum at baseline with data post-randomization, 1 evaluable PK blood sample (OZ439/FQ) post dose, adequate documentation of dosing & sampling date, without any major protocol deviation related to drug administration (e.g. vomiting after drug intake). Here,"overall number of participants analyzed"=participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ferroquine 400 mg | Ferroquine 400 mg + Artefenomel 300 mg | Ferroquine 400 mg + Artefenomel 600 mg | Ferroquine 400 mg + Artefenomel 1000 mg
Number analyzed (Participants) | 26 | 31 | 33 | 31
percentage of participants | 80.8 [62.1 to 91.5] | 90.3 [75.1 to 96.7] | 90.9 [76.4 to 96.9] | 87.1 [71.1 to 94.9]

2. Secondary Outcome: Percentage of Participants With Crude Adequate Clinical and Parasitological Response at Day 28
Description: ACPR: absence of parasitemia at Day 28, irrespective of AT, in participants not meeting any criteria of ETF: DS/SoC/SM at Day 1, 2 or 3 in presence of parasitemia, concomitant to at least 1 positive parasitemia; or parasitemia on Day 2 > Day 0 irrespective of AT; or parasitemia on Day 3 with AT >=37.5°C; or parasitemia count on Day 3 >=25% on Day 0, or LCF: DS/SM in presence of parasitemia between Day 4 and 28, concomitant to at least one positive parasitemia; or presence of parasitemia and AT>=37.5°C on Day 4 to Day 28, or LPF: presence of parasitemia between Day 7 and 28 and AT<37.5°C or having rescue therapy for malaria. PCR-corrected ACPR applied to recrudescence (appearance of asexual parasites after clearance of initial infection with genotype identical to that present at Baseline), excluding participants with re-infection, whereas crude ACPR does not distinguish reinfection (new clone of parasite) or recrudescence.
Time Frame: Day 28
Population: Analysis was performed on PK/PD efficacy population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ferroquine 400 mg | Ferroquine 400 mg + Artefenomel 300 mg | Ferroquine 400 mg + Artefenomel 600 mg | Ferroquine 400 mg + Artefenomel 1000 mg
Number analyzed (Participants) | 31 | 33 | 36 | 32
percentage of participants | 64.5 [46.9 to 78.9] | 81.8 [65.6 to 91.4] | 77.8 [61.9 to 88.3] | 78.1 [61.2 to 89]

3. Secondary Outcome: Parasitemia: Change From Baseline in Number of Parasites Per Microliter of Blood at 6, 12, 18, 24, 30, 36, 48, 72, 96, 120, 144 and 168 Hours
Description: Parasitemia (quantitative content of parasites present in the blood) at baseline until Day 7 (i.e. 168 hours) was assessed by optical microscope.
Time Frame: Baseline, 6, 12, 18, 24, 30, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
Population: Analysis was performed on modified intention-to-treat (mITT) population which included all randomized participants with parasitological confirmed P.falciparum malaria at baseline with parasitemia data post-randomization, received the single administration of OZ439/FQ. Here, "number analyzed" = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: parasites per microliter
Arm/Group | Ferroquine 400 mg | Ferroquine 400 mg + Artefenomel 300 mg | Ferroquine 400 mg + Artefenomel 600 mg | Ferroquine 400 mg + Artefenomel 1000 mg
Number analyzed (Participants) | 35 | 36 | 36 | 33
parasites per microliter
  Baseline | 17496.0 (11889.55) | 18799.6 (13559.14) | 15171.9 (13012.53) | 20546.8 (13835.31)
  Change from baseline at 6 hours post-dose: number analyzed (Participants) | 35 | 36 | 36 | 32
  Change from baseline at 6 hours post-dose | -1349.3 (11331.78) | -96.9 (11699.28) | 8515.4 (44264.14) | 893.2 (21052.27)
  Change from baseline at 12 hours post-dose: number analyzed (Participants) | 35 | 36 | 35 | 33
  Change from baseline at 12 hours post-dose | -5721.5 (12441.39) | -11471.6 (13399.27) | -4156.6 (34663.71) | -11319.4 (15490.43)
  Change from baseline at 18 hours post-dose: number analyzed (Participants) | 34 | 36 | 36 | 33
  Change from baseline at 18 hours post-dose | -9181.2 (11892.89) | -17021.4 (13015.29) | -9447.5 (32303.36) | -18281.9 (13796.37)
  Change from baseline at 24 hours post-dose: number analyzed (Participants) | 34 | 36 | 36 | 33
  Change from baseline at 24 hours post-dose | -14238.4 (11402.25) | -17939.0 (13061.86) | -10674.6 (29868.45) | -19461.9 (14049.02)
  Change from baseline at 30 hours post-dose: number analyzed (Participants) | 34 | 35 | 36 | 32
  Change from baseline at 30 hours post-dose | -16571.1 (12354.88) | -19110.5 (13556.35) | -13299.6 (17452.15) | -19657.5 (14393.75)
  Change from baseline at 36 hours post-dose: number analyzed (Participants) | 34 | 36 | 36 | 33
  Change from baseline at 36 hours post-dose | -17036.9 (12307.57) | -18792.2 (13548.16) | -14573.9 (13623.86) | -19587.9 (14051.82)
  Change from baseline at 48 hours post-dose: number analyzed (Participants) | 34 | 36 | 36 | 33
  Change from baseline at 48 hours post-dose | -17595.3 (12037.99) | -17706.1 (13389.25) | -14542.3 (13547.11) | -20327.7 (13739.17)
  Change from baseline at 72 hours post-dose: number analyzed (Participants) | 33 | 35 | 34 | 32
  Change from baseline at 72 hours post-dose | -18231.8 (11801.65) | -18396.3 (13091.47) | -15333.7 (13382.41) | -20314.2 (13980.12)
  Change from baseline at 96 hours post-dose: number analyzed (Participants) | 31 | 33 | 35 | 31
  Change from baseline at 96 hours post-dose | -18287.6 (12011.77) | -19024.7 (13200.22) | -15258.5 (13191.95) | -20662.0 (14108.54)
  Change from baseline at 120 hours post-dose: number analyzed (Participants) | 29 | 33 | 35 | 32
  Change from baseline at 120 hours post-dose | -19280.0 (12145.86) | -19024.7 (13200.22) | -15265.3 (13190.14) | -20350.4 (14010.21)
  Change from baseline at 144 hours post-dose: number analyzed (Participants) | 32 | 33 | 35 | 31
  Change from baseline at 144 hours post-dose | -18526.0 (11889.52) | -19023.3 (13198.28) | -15254.5 (13190.39) | -20029.7 (14121.74)
  Change from baseline at 168 hours post-dose: number analyzed (Participants) | 31 | 31 | 34 | 32
  Change from baseline at 168 hours post-dose | -18962.8 (11813.20) | -18922.2 (13141.19) | -15268.5 (13388.49) | -20349.5 (14010.98)

4. Secondary Outcome: Observed Parasite Reduction Ratio (PRR) at 24 Hours, 48 Hours, and 72 Hours
Description: The observed PRR was defined as the ratio of the number of parasites at time t=0 (baseline) divided by the parasite count at each specified time t (post-treatment). If the post dose parasite count = 0 (due to a negative parasitemia) then a value of 1 parasite per microliter was imputed to allow a parasite reduction ratio calculation.
Time Frame: Baseline, 24, 48 and 72 hours post-dose
Population: Analysis was performed on mITT population. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Ferroquine 400 mg | Ferroquine 400 mg + Artefenomel 300 mg | Ferroquine 400 mg + Artefenomel 600 mg | Ferroquine 400 mg + Artefenomel 1000 mg
Number analyzed (Participants) | 35 | 36 | 36 | 33
ratio
  At Hour 24: number analyzed (Participants) | 34 | 36 | 36 | 33
  At Hour 24 | 638.436 (2013.8609) | 5921.197 (11566.1520) | 5715.046 (9364.8892) | 7929.720 (12675.8348)
  At Hour 48: number analyzed (Participants) | 34 | 36 | 36 | 33
  At Hour 48 | 9709.093 (13987.7127) | 17594.700 (13521.9507) | 13120.409 (13182.3022) | 19328.057 (14392.7604)
  At Hour 72: number analyzed (Participants) | 33 | 35 | 35 | 32
  At Hour 72 | 15655.447 (12806.4644) | 18069.583 (13409.1341) | 14561.409 (13657.0665) | 19125.715 (14516.8397)

5. Secondary Outcome: Time to 50% and 99% Parasite Reduction
Description: Time to 50% and 99% parasite reduction was defined as time needed for the parasitemia (quantitative content of parasites present in blood) to be reduced to 50% and 99% of the initial value, respectively.
Time Frame: Up to Day 28
Population: Analysis was performed on mITT population. Here, "Overall Number of Participants Analyzed" = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Ferroquine 400 mg | Ferroquine 400 mg + Artefenomel 300 mg | Ferroquine 400 mg + Artefenomel 600 mg | Ferroquine 400 mg + Artefenomel 1000 mg
Number analyzed (Participants) | 21 | 28 | 28 | 25
hours
  Time to 50% Parasite reduction | 14.07 (5.604) | 7.74 (4.636) | 7.78 (3.786) | 9.47 (7.976)
  Time to 99% Parasite reduction | 36.92 (9.988) | 19.33 (6.107) | 18.34 (5.523) | 22.95 (17.069)

6. Secondary Outcome: Parasite Clearance Time (PCT)
Description: PCT was defined as the time (in hours) from the start of study drug administration until the time of first negative blood film (no asexual parasites by microscopy). This first negative film was confirmed by a second negative film which was taken >=6 to <=12 hours of the first film. If the second film was performed <6 hours or >12 hours of the first film, then the parasite clearance was confirmed or invalidated by the third (thick) film following the second one, whatever the timing of this third film: If the third film was negative, then the clearance was considered confirmed and if the third film was positive, then the clearance was invalidated. Kaplan-Meier method was used for the estimation.
Time Frame: From the start of study drug administration up to the time of the first negative blood film (up to Day 28)
Population: Analysis was performed on mITT population.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Ferroquine 400 mg | Ferroquine 400 mg + Artefenomel 300 mg | Ferroquine 400 mg + Artefenomel 600 mg | Ferroquine 400 mg + Artefenomel 1000 mg
Number analyzed (Participants) | 35 | 36 | 36 | 33
hours | 56.1 [48.0 to 72.0] | 30.0 [30.0 to 30.0] | 30.0 [24.1 to 30.1] | 30.0 [24.0 to 30.0]

7. Secondary Outcome: Parasite Clearance Rate
Description: Parasite clearance rate (k) is the minus slope of the natural logarithm parasitemia versus time linear relationship, after exclusion of outliers, lag phase and Tail, using the worldwide antimalarial resistance network, Parasite Clearance Estimator.
Time Frame: Up to Day 28
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: 1 per hour
Arm/Group | Ferroquine 400 mg | Ferroquine 400 mg + Artefenomel 300 mg | Ferroquine 400 mg + Artefenomel 600 mg | Ferroquine 400 mg + Artefenomel 1000 mg
Number analyzed (Participants) | 21 | 28 | 28 | 25
1 per hour | 0.1956 (0.07627) | 0.3609 (0.09963) | 0.3962 (0.11983) | 0.3581 (0.12484)

8. Secondary Outcome: Time to Re-emergence
Description: Time to re-emergence (in days) was defined as the time to appearance of asexual parasites after clearance of initial infection irrespective of genotype. Re-emergence was confirmed by microscopy (positive blood smear). Participants with confirmed parasite clearance were included in the analysis and Kaplan-Meier method was used for estimation.
Time Frame: Up to Day 28
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Ferroquine 400 mg | Ferroquine 400 mg + Artefenomel 300 mg | Ferroquine 400 mg + Artefenomel 600 mg | Ferroquine 400 mg + Artefenomel 1000 mg
Number analyzed (Participants) | 32 | 35 | 34 | 32
days | NA [28.0 to NA] — Median and upper limit of confidence interval (CI) was not estimable due to very low number of participants with events. | NA [NA to NA] — Median and 95% CI was not estimable due to very low number of participants with the events . | NA [NA to NA] — Median and 95% CI was not estimable due to very low number of participants with the events . | NA [NA to NA] — Median and 95% CI was not estimable due to very low number of participants with the events .

9. Secondary Outcome: Time to Recrudescence
Description: Time to recrudescence (in days) was defined as the time to appearance of asexual parasites after clearance of initial infection with a genotype identical to that of parasites present at Baseline. Recrudescence was confirmed by PCR analysis. Participants with confirmed parasite clearance were included in the analysis and Kaplan-Meier method was used for estimation.
Time Frame: Up to Day 28
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Ferroquine 400 mg | Ferroquine 400 mg + Artefenomel 300 mg | Ferroquine 400 mg + Artefenomel 600 mg | Ferroquine 400 mg + Artefenomel 1000 mg
Number analyzed (Participants) | 32 | 35 | 34 | 32
days | NA [NA to NA] — Median and 95% CI was not estimable due to very low number of participants with the events. | NA [NA to NA] — Median and 95% CI was not estimable due to very low number of participants with the events. | NA [NA to NA] — Median and 95% CI was not estimable due to very low number of participants with the events. | NA [NA to NA] — Median and 95% CI was not estimable due to very low number of participants with the events.

10. Secondary Outcome: Time to Re-infection
Description: Time to re-infection (in days) was defined as the time to appearance of asexual parasites after clearance of initial infection with a genotype that differed from that of parasites present at Baseline. Re-infection was confirmed by PCR analysis. Participants with confirmed parasite clearance were involved in the analysis and Kaplan-Maier method was used for estimation.
Time Frame: Up to Day 28
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Ferroquine 400 mg | Ferroquine 400 mg + Artefenomel 300 mg | Ferroquine 400 mg + Artefenomel 600 mg | Ferroquine 400 mg + Artefenomel 1000 mg
Number analyzed (Participants) | 32 | 35 | 34 | 32
days | NA [NA to NA] — Median and 95% CI was not estimable due to very low number of participants with the events. | NA [NA to NA] — Median and 95% CI was not estimable due to very low number of participants with the events. | NA [NA to NA] — Median and 95% CI was not estimable due to very low number of participants with the events. | NA [NA to NA] — Median and 95% CI was not estimable due to very low number of participants with the events.

11. Secondary Outcome: Time Elapsed Below the Limit of Quantification (LOQ) of Parasitemia
Description: The time elapsed below LOQ (LOQ expressed in parasites/microliter) of parasitemia (quantitative content of parasites present in the blood) was defined as the time (in days) for which no parasites were seen i.e., time corresponding to PCT, up to the time of occurrence of a new malaria infection or recrudescence. If there was no occurrence of a new malaria infection or recrudescence, then this was the time corresponding to the first negative thick blood film, until the end of study. PCT (k) is the minus slope of the natural logarithm parasitemia versus time linear relationship, after exclusion of outliers, lag phase and Tail, using the worldwide antimalarial resistance network, Parasite clearance estimator. Participants with confirmed parasite clearance were involved in the analysis and Kaplan-Meier method was used for estimation.
Time Frame: Up to Day 28
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Ferroquine 400 mg | Ferroquine 400 mg + Artefenomel 300 mg | Ferroquine 400 mg + Artefenomel 600 mg | Ferroquine 400 mg + Artefenomel 1000 mg
Number analyzed (Participants) | 32 | 35 | 34 | 32
days | 25.0 [23.0 to 26.0] | 26.0 [26.0 to 27.0] | 26.5 [26.0 to 27.0] | 26.0 [26.0 to 27.0]

12. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs) and Adverse Event of Special Interest (AESI)
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug and did not necessarily had to have a causal relationship with the treatment. SAEs were any untoward medical occurrence that resulted in any of the following outcomes: death, life-threatening, required initial or prolonged in-patient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event. TEAEs were defined as AEs that developed or worsened or became serious during on-treatment phase that was defined as the time from the start of study drug up to the Day 28. AE of special interest (AESI) was an AE (serious or non-serious) of scientific and medical concern specific to the Sponsor's product or program, for which ongoing monitoring and immediate notification by the Investigator to the Sponsor was required.
Time Frame: From Baseline up to Day 28
Population: Analysis was performed on safety population: participants who received single administration of OZ439/FQ and were analyzed according to the treatment actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Ferroquine 400 mg | Ferroquine 400 mg + Artefenomel 300 mg | Ferroquine 400 mg + Artefenomel 600 mg | Ferroquine 400 mg + Artefenomel 1000 mg
Number analyzed (Participants) | 35 | 36 | 36 | 33
Participants
  Any TEAE | 18 | 21 | 24 | 24
  Any treatment-emergent SAE | 0 | 0 | 1 | 0
  Any treatment-emergent AESI | 0 | 1 | 0 | 1
  Any TEAE led to treatment discontinuation | 0 | 0 | 0 | 0
  Any TEAE led to death | 0 | 0 | 0 | 0

13. Secondary Outcome: Pharmacokinetics (PK): Concentration of OZ439 in Plasma
Description: Concentrations of OZ439 in plasma was analyzed by liquid chromatography tandem mass spectroscopy (LC-MS/MS). The lower limit of quantification (LLOQ) was 1 nanograms per milliliter for analysis of OZ439. Data for this outcome measure was not planned to be collected and analyzed for "Ferroquine 400 mg" arm, since artefenomel was not administered.
Time Frame: 1, 2, 4, 6, 12, 24, 48, 72, 120, 168 and 336 hours post-dose
Population: Analysis was performed on PK population which included all participants who received OZ439 and had at least one evaluable blood sample for PK OZ439 post study drug administration and with adequate documentation of date of dosing and date of sampling. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter
Arm/Group | Ferroquine 400 mg + Artefenomel 300 mg | Ferroquine 400 mg + Artefenomel 600 mg | Ferroquine 400 mg + Artefenomel 1000 mg
Number analyzed (Participants) | 36 | 36 | 33
nanograms per milliliter
  1 hour post-dose: number analyzed (Participants) | 35 | 35 | 32
  1 hour post-dose | 88.641 (104.631) | 149.199 (87.153) | 188.423 (82.588)
  2 hours post-dose: number analyzed (Participants) | 35 | 34 | 32
  2 hours post-dose | 269.075 (59.803) | 450.218 (58.642) | 655.851 (58.311)
  4 hours post-dose: number analyzed (Participants) | 35 | 35 | 32
  4 hours post-dose | 349.134 (54.880) | 576.673 (54.357) | 978.649 (60.263)
  6 hours post-dose: number analyzed (Participants) | 35 | 35 | 32
  6 hours post-dose | 234.375 (52.902) | 478.929 (87.523) | 865.581 (75.154)
  12 hours post-dose: number analyzed (Participants) | 34 | 35 | 32
  12 hours post-dose | 92.614 (60.229) | 164.028 (99.433) | 369.335 (85.243)
  24 hours post-dose: number analyzed (Participants) | 33 | 33 | 31
  24 hours post-dose | 17.526 (65.757) | 48.257 (107.605) | 84.167 (78.221)
  48 hours post-dose: number analyzed (Participants) | 33 | 33 | 32
  48 hours post-dose | 6.097 (54.492) | 14.611 (95.627) | 29.554 (83.028)
  72 hours post-dose: number analyzed (Participants) | 32 | 33 | 30
  72 hours post-dose | 3.224 (50.406) | 8.162 (77.493) | 16.665 (83.936)
  120 hours post-dose: number analyzed (Participants) | 25 | 32 | 30
  120 hours post-dose | 2.144 (39.859) | 5.339 (61.816) | 8.596 (77.245)
  168 hours post-dose: number analyzed (Participants) | 21 | 32 | 30
  168 hours post-dose | 1.745 (38.466) | 3.408 (73.232) | 5.903 (78.608)
  336 hours post-dose: number analyzed (Participants) | 6 | 21 | 25
  336 hours post-dose | 1.227 (19.402) | 1.970 (66.212) | 3.149 (58.029)

14. Secondary Outcome: Pharmacokinetics: Concentration of FQ and Its Active Metabolite SSR97213 in Blood
Description: Concentrations of FQ and SSR97213 in blood was analyzed by LC-MS/MS. The LLOQ was 5 nanograms per milliliter for analysis of FQ and SSR97213.
Time Frame: 1, 4, 6, 8, 12, 24, 72, 168, 336 and 672 hours post-dose
Population: Analysis was performed on PK population which included all participants who received FQ and had at least one evaluable blood sample for PK FQ post study drug administration and with adequate documentation of date of dosing and date of sampling. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter
Arm/Group | Ferroquine 400 mg | Ferroquine 400 mg + Artefenomel 300 mg | Ferroquine 400 mg + Artefenomel 600 mg | Ferroquine 400 mg + Artefenomel 1000 mg
Number analyzed (Participants) | 35 | 36 | 36 | 33
nanograms per milliliter
  1 hour post-dose: FQ: number analyzed (Participants) | 32 | 33 | 25 | 25
  1 hour post-dose: FQ | 36.094 (80.476) | 27.214 (79.000) | 21.165 (55.491) | 26.599 (95.999)
  1 hour post-dose: SSR97213: number analyzed (Participants) | 8 | 2 | 2 | 2
  1 hour post-dose: SSR97213 | 13.209 (54.030) | 10.375 (15.713) | 6.161 (9.504) | 6.805 (28.203)
  4 hours post-dose: FQ: number analyzed (Participants) | 35 | 35 | 35 | 31
  4 hours post-dose: FQ | 64.934 (87.235) | 100.569 (61.578) | 79.656 (74.707) | 97.007 (72.230)
  4 hours post-dose: SSR97213: number analyzed (Participants) | 27 | 27 | 29 | 26
  4 hours post-dose: SSR97213 | 20.079 (90.358) | 29.632 (49.701) | 18.377 (98.310) | 17.559 (68.694)
  6 hours post-dose: FQ: number analyzed (Participants) | 35 | 35 | 35 | 32
  6 hours post-dose: FQ | 69.005 (75.045) | 92.657 (50.449) | 84.803 (75.544) | 95.062 (126.388)
  6 hours post-dose: SSR97213: number analyzed (Participants) | 30 | 30 | 29 | 28
  6 hours post-dose: SSR97213 | 23.170 (82.875) | 28.098 (53.438) | 25.954 (88.481) | 20.687 (70.211)
  8 hours post-dose: FQ: number analyzed (Participants) | 34 | 35 | 35 | 32
  8 hours post-dose: FQ | 64.293 (70.724) | 82.639 (49.891) | 78.196 (72.454) | 82.990 (69.989)
  8 hours post-dose: SSR97213: number analyzed (Participants) | 29 | 29 | 29 | 29
  8 hours post-dose: SSR97213 | 25.131 (66.944) | 29.319 (48.679) | 25.304 (78.822) | 20.299 (63.388)
  12 hours post-dose: FQ: number analyzed (Participants) | 35 | 35 | 35 | 32
  12 hours post-dose: FQ | 50.621 (57.540) | 68.384 (50.887) | 59.106 (70.461) | 71.743 (61.238)
  12 hours post-dose: SSR97213: number analyzed (Participants) | 31 | 31 | 30 | 31
  12 hours post-dose: SSR97213 | 19.957 (61.856) | 24.385 (48.408) | 20.615 (77.739) | 18.203 (64.197)
  24 hours post-dose: FQ: number analyzed (Participants) | 34 | 36 | 35 | 32
  24 hours post-dose: FQ | 44.351 (52.316) | 53.211 (48.834) | 47.568 (61.373) | 51.250 (75.940)
  24 hours post-dose: SSR97213: number analyzed (Participants) | 32 | 33 | 30 | 31
  24 hours post-dose: SSR97213 | 18.874 (56.412) | 22.967 (55.037) | 19.826 (70.907) | 16.763 (69.091)
  72 hours post-dose: FQ: number analyzed (Participants) | 34 | 35 | 35 | 31
  72 hours post-dose: FQ | 25.343 (35.315) | 31.161 (47.829) | 31.373 (70.287) | 29.792 (76.912)
  72 hours post-dose: SSR97213: number analyzed (Participants) | 32 | 33 | 30 | 29
  72 hours post-dose: SSR97213 | 16.757 (46.038) | 20.059 (45.134) | 21.315 (68.366) | 17.756 (82.612)
  168 hours post-dose: FQ: number analyzed (Participants) | 31 | 31 | 34 | 31
  168 hours post-dose: FQ | 16.973 (39.627) | 20.524 (39.625) | 21.543 (63.679) | 21.322 (62.951)
  168 hours post-dose: SSR97213: number analyzed (Participants) | 31 | 30 | 31 | 30
  168 hours post-dose: SSR97213 | 16.308 (52.300) | 19.196 (46.115) | 20.463 (55.587) | 19.108 (62.123)
  336 hours post-dose: FQ: number analyzed (Participants) | 28 | 31 | 31 | 29
  336 hours post-dose: FQ | 10.543 (36.770) | 11.678 (38.490) | 12.469 (48.236) | 11.263 (82.611)
  336 hours post-dose: SSR97213: number analyzed (Participants) | 31 | 31 | 31 | 30
  336 hours post-dose: SSR97213 | 13.612 (45.485) | 14.797 (46.036) | 15.647 (47.974) | 13.686 (72.213)
  672 hours post-dose: FQ: number analyzed (Participants) | 11 | 17 | 20 | 21
  672 hours post-dose: FQ | 6.737 (18.832) | 7.623 (28.348) | 7.601 (29.047) | 7.342 (53.998)
  672 hours post-dose: SSR97213: number analyzed (Participants) | 26 | 30 | 28 | 25
  672 hours post-dose: SSR97213 | 9.751 (41.862) | 10.324 (33.482) | 10.977 (34.251) | 12.014 (59.403)

15. Secondary Outcome: Pharmacokinetics: Maximum Observed Plasma Concentration (Cmax) of Artefenomel
Description: Cmax is the maximum observed plasma concentration of Artefenomel. Data for this outcome measure was not planned to be collected and analyzed for "Ferroquine 400 mg" arm, since artefenomel was not administered.
Time Frame: Pre-dose, 1, 2, 4, 6, 12, 24, 48, 72, 120, 168 and 336 hours post-dose
Population: Analysis was performed on PK/PD efficacy population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter
Arm/Group | Ferroquine 400 mg + Artefenomel 300 mg | Ferroquine 400 mg + Artefenomel 600 mg | Ferroquine 400 mg + Artefenomel 1000 mg
Number analyzed (Participants) | 33 | 36 | 32
nanograms per milliliter | 277.3 (169) | 488.3 (232) | 920.6 (77)

16. Secondary Outcome: Pharmacokinetics: Time to Reach Maximum Plasma Concentration (Tmax) of Artefenomel
Description: tmax is the time taken by the drug to reach the maximum plasma concentration. Data for this outcome measure was not planned to be collected and analyzed for "Ferroquine 400 mg" arm, since artefenomel was not administered.
Time Frame: Pre-dose, 1, 2, 4, 6, 12, 24, 48, 72, 120, 168 and 336 hours post-dose
Population: Focus of PK assessment was to support the analysis of exposure versus efficacy relationship (PK and PD). Since tmax was not considered relevant to the objective of exposure-response analysis, data for this outcome measure were not collected and reported.
Arm/Group | Ferroquine 400 mg + Artefenomel 300 mg | Ferroquine 400 mg + Artefenomel 600 mg | Ferroquine 400 mg + Artefenomel 1000 mg
Number analyzed (Participants) | 0 | 0 | 0

17. Secondary Outcome: Pharmacokinetics: Plasma Concentration at 168 Hours Post-dose (C168h) of Artefenomel
Description: The observed plasma concentration of artefenomel post 168 hours of drug administration. Data for this outcome measure was not planned to be collected and analyzed for "Ferroquine 400 mg" arm, since artefenomel was not administered.
Time Frame: At 168 hours post-dose
Population: Analysis was performed on PK/PD efficacy population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter
Arm/Group | Ferroquine 400 mg + Artefenomel 300 mg | Ferroquine 400 mg + Artefenomel 600 mg | Ferroquine 400 mg + Artefenomel 1000 mg
Number analyzed (Participants) | 33 | 36 | 32
nanograms per milliliter | 0.9251 (110) | 2.152 (202) | 4.445 (165)

18. Secondary Outcome: Pharmacokinetics: Area Under the Concentration Curve (AUC) Form Time 0 to Infinity (AUC0-inf]) of Artefenomel
Description: Area under the plasma concentration versus time curve from time 0 to infinity. Data for this outcome measure was not planned to be collected and analyzed for "Ferroquine 400 mg" arm, since artefenomel was not administered.
Time Frame: Pre-dose, 1, 2, 4, 6, 12, 24, 48, 72, 120, 168 and 336 hours post-dose
Population: Analysis was performed on PK/PD efficacy population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*hour per milliliter
Arm/Group | Ferroquine 400 mg + Artefenomel 300 mg | Ferroquine 400 mg + Artefenomel 600 mg | Ferroquine 400 mg + Artefenomel 1000 mg
Number analyzed (Participants) | 33 | 36 | 32
micrograms*hour per milliliter | 3.269 (113) | 6.46 (181) | 13.05 (114)

19. Secondary Outcome: Pharmacokinetics: Terminal Half-life (t1/2) of Artefenomel
Description: Terminal t1/2 is defined as the time required for the plasma concentration of a drug to decrease by half of its initial concentration. Data for this outcome measure was not planned to be collected and analyzed for "Ferroquine 400 mg" arm, since artefenomel was not administered.
Time Frame: Pre-dose, 1, 2, 4, 6, 12, 24, 48, 72, 120, 168 and 336 hours post-dose
Population: Focus of PK assessment was to support the analysis of exposure versus efficacy relationship (PK and PD). Since terminal t1/2 was not considered relevant to the objective of exposure-response analysis, therefore data for this outcome measure were not collected and reported.
Arm/Group | Ferroquine 400 mg + Artefenomel 300 mg | Ferroquine 400 mg + Artefenomel 600 mg | Ferroquine 400 mg + Artefenomel 1000 mg
Number analyzed (Participants) | 0 | 0 | 0

20. Secondary Outcome: Pharmacokinetics: Maximum Observed Plasma Concentration of Ferroquine and Its Active Metabolite SSR97213
Description: Cmax is the maximum observed plasma concentration of Ferroquine.
Time Frame: Pre-dose, 1, 4, 6, 8, 12, 24, 72, 168, 336 and 672 hours post-dose
Population: Analysis was performed on PK/PD efficacy population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter
Arm/Group | Ferroquine 400 mg | Ferroquine 400 mg + Artefenomel 300 mg | Ferroquine 400 mg + Artefenomel 600 mg | Ferroquine 400 mg + Artefenomel 1000 mg
Number analyzed (Participants) | 31 | 33 | 36 | 32
nanograms per milliliter
  FQ | 80.99 (61) | 79.95 (93) | 72.64 (88) | 82.45 (95)
  SSR97213 | 24.58 (61) | 22.65 (83) | 19.14 (99) | 19.76 (78)

21. Secondary Outcome: Pharmacokinetics: Time to Reach Maximum Plasma Concentration of Ferroquine and Its Active Metabolite SSR97213
Description: tmax is the time taken by the drug to reach the maximum plasma concentration.
Time Frame: Pre-dose, 1, 4, 6, 8, 12, 24, 72, 168, 336 and 672 hours post-dose
Population: Focus of PK assessment was to support the analysis of exposure versus efficacy relationship (PK and PD). Since tmax was not considered relevant to the objective of exposure-response analysis, therefore data for this outcome measure were not collected and reported.
Arm/Group | Ferroquine 400 mg | Ferroquine 400 mg + Artefenomel 300 mg | Ferroquine 400 mg + Artefenomel 600 mg | Ferroquine 400 mg + Artefenomel 1000 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

22. Secondary Outcome: Pharmacokinetics: Plasma Concentration at 168 Hours Post-dose of Ferroquine and Its Active Metabolite SSR97213
Description: The observed plasma concentration of FQ and SSR97213 post 168 hours of FQ administration.
Time Frame: At 168 hours post-dose
Population: Analysis was performed on PK/PD efficacy population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter
Arm/Group | Ferroquine 400 mg | Ferroquine 400 mg + Artefenomel 300 mg | Ferroquine 400 mg + Artefenomel 600 mg | Ferroquine 400 mg + Artefenomel 1000 mg
Number analyzed (Participants) | 31 | 33 | 36 | 32
nanograms per milliliter
  FQ | 15.86 (44) | 18.32 (42) | 18.69 (52) | 17.83 (60)
  SSR97213 | 16.15 (51) | 16.03 (68) | 15.2 (78) | 14.95 (86)

23. Secondary Outcome: Pharmacokinetics: Area Under the Concentration Curve Form Time 0 to Day 28 (AUC0-28) of Ferroquine and Its Active Metabolite SSR97213
Description: Area under the plasma concentration versus time curve from time 0 to Day 28 (i.e. 672 hours).
Time Frame: Pre-dose, 1, 4, 6, 8, 12, 24, 72, 168, 336 and 672 hours post-dose
Population: Analysis was performed on PK/PD efficacy population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*hour per milliliter
Arm/Group | Ferroquine 400 mg | Ferroquine 400 mg + Artefenomel 300 mg | Ferroquine 400 mg + Artefenomel 600 mg | Ferroquine 400 mg + Artefenomel 1000 mg
Number analyzed (Participants) | 31 | 33 | 36 | 32
micrograms*hour per milliliter
  FQ | 8.874 (42) | 10.33 (40) | 10.13 (51) | 10.14 (56)
  SSR97213 | 8.878 (48) | 9.051 (56) | 8.483 (68) | 8.487 (71)

24. Secondary Outcome: Pharmacokinetics: Area Under the Concentration Curve From Time 0 to Infinity of Ferroquine and Its Active Metabolite SSR97213
Description: Area under the plasma concentration versus time curve from time 0 to infinity.
Time Frame: Pre-dose, 1, 4, 6, 8, 12, 24, 72, 168, 336 and 672 hours post-dose
Population: Analysis was performed on PK/PD efficacy population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*hour per milliliter
Arm/Group | Ferroquine 400 mg | Ferroquine 400 mg + Artefenomel 300 mg | Ferroquine 400 mg + Artefenomel 600 mg | Ferroquine 400 mg + Artefenomel 1000 mg
Number analyzed (Participants) | 31 | 33 | 36 | 32
micrograms*hour per milliliter
  FQ | 15.5 (47) | 17.81 (43) | 16.3 (63) | 16.87 (59)
  SSR97213 | 19.58 (53) | 20.09 (48) | 17.94 (69) | 18.32 (68)

25. Secondary Outcome: Pharmacokinetics: Terminal Half-life of Ferroquine
Description: Terminal t1/2 is defined as the time required for the plasma concentration of a drug to decrease by half of its initial concentration.
Time Frame: Pre-dose, 1, 4, 6, 8, 12, 24, 72, 168, 336 and 672 hours post-dose
Population: as for outcome 19
Arm/Group | Ferroquine 400 mg | Ferroquine 400 mg + Artefenomel 300 mg | Ferroquine 400 mg + Artefenomel 600 mg | Ferroquine 400 mg + Artefenomel 1000 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From Baseline up to Day 28
Description: Reported AEs were TEAEs, defined as AEs that developed/worsened or became serious during on-treatment phase - defined as the time from the start of the first dose of study drug administration up to Day 28. Analysis was performed on safety population.
Arm/Group | Ferroquine 400 mg | Ferroquine 400 mg + Artefenomel 300 mg | Ferroquine 400 mg + Artefenomel 600 mg | Ferroquine 400 mg + Artefenomel 1000 mg
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/36 | 0/36 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/36 | 1/36 | 0/33
Other Adverse Events (participants affected / at risk) | 13/35 | 17/36 | 17/36 | 22/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ferroquine 400 mg (N=35) | Ferroquine 400 mg + Artefenomel 300 mg (N=36) | Ferroquine 400 mg + Artefenomel 600 mg (N=36) | Ferroquine 400 mg + Artefenomel 1000 mg (N=33)
Malaria (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ferroquine 400 mg (N=35) | Ferroquine 400 mg + Artefenomel 300 mg (N=36) | Ferroquine 400 mg + Artefenomel 600 mg (N=36) | Ferroquine 400 mg + Artefenomel 1000 mg (N=33)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 4 (4) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (3) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (3) | 3 (3) | 5 (5) | 10 (10)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 1 (1) | 4 (4)
Malaria (Infections and infestations) | 7 (7) | 6 (6) | 7 (7) | 6 (6)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 2 (3)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
Headache (Nervous system disorders) | 3 (3) | 6 (10) | 1 (1) | 7 (9)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2017-11-13): https://cdn.clinicaltrials.gov/large-docs/39/NCT03660839/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-29): https://cdn.clinicaltrials.gov/large-docs/39/NCT03660839/SAP_001.pdf